CLINICAL TRIAL: NCT03589326
Title: A Phase 3, Randomized, Open-label, Multicenter Study Comparing Ponatinib Versus Imatinib, Administered in Combination With Reduced-Intensity Chemotherapy, in Patients With Newly Diagnosed Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL)
Brief Title: A Study of Ponatinib Versus Imatinib in Adults With Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ponatinib-3001; U1111-1206-2370 (Other: World Health Organization); HC6-24-c220300 (Registry Identifier: Health Canada); jRCT2031210230 (Registry Identifier: jRCT); 2023-508463-71-00 (EU CTIS Number)
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ALL)
Keywords: Ponatinib; Imatinib mesylate; Bcr-Abl Tyrosine Kinase; Bcr-abl fusion proteins; Iclusig; Gleevec
MeSH Terms: interventions — ponatinib; Imatinib Mesylate; Vincristine; Dexamethasone; Cytarabine; Methotrexate; Prednisone

STUDY DESIGN:
Masking Description: It is an open-label trial, therefore investigators and participants are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Ponatinib 30 milligram (mg) (Experimental): Ponatinib 30 mg, tablets, orally, once daily (QD), with vincristine 1.4 mg/m^2 (max 2 mg) intravenous (IV), on Days 1 and 14 and dexamethasone 40 mg (<60 years [yrs]) and 20 mg (≥60 yrs), orally, once on Days 1 to 4, Days 11 to 14 for up to 3 cycles (each cycle=28 days) in induction phase (reduced dose of ponatinib 15 mg upon achievement of MRD-negative CR at end of induction) followed by ponatinib last induction phase dose with cytarabine, 1000 mg/m^2 as 2-hour IV infusion (<60 yrs) and 250 mg/m^2 (≥60 yrs) every 12 hours, IV on Days 1, 3, 5 of Cycles 2,4,6 and methotrexate, 1000 mg/m^2 (<60 yrs) and 250 mg/m^2 (≥60 yrs), IV infusion, on Day 1 of cycles 1, 3, 5 in consolidation phase followed by ponatinib last consolidation phase dose with vincristine 1.4 mg/m^2 (max 2 mg), IV, on Day 1 and prednisone 200 mg (<60 yrs), 100 mg (≥60-69 yrs) and 50 mg(≥70 yrs) on Days 1 to 5 for up to 11 cycles in maintenance phase up to data cut-off date: 12 August 2022.
  Interventions: Drug: Ponatinib; Drug: Vincristine; Drug: Dexamethasone; Drug: Cytarabine; Drug: Methotrexate; Drug: Prednisone
- Cohort B: Imatinib 600 mg (Active Comparator): Imatinib 600 mg, tablets, orally, QD, with vincristine 1.4 mg/m^2 (max 2 mg), IV, on Days 1 and 14 and dexamethasone 40 mg (<60 yrs) and 20 mg (≥60 yrs), orally, once on Days 1 to 4 and Days 11 to 14 in each 28-day cycle for up to 3 cycles in the induction phase followed by imatinib 600 mg, tablets, orally, QD, with cytarabine, 1000 mg/m^2 every 12 hours as a 2-hour-IV infusion (<60 yrs) and 250 mg/m^2 every 12 hours (≥60 yrs), IV on Days 1, 3, and 5 of each 28-day even cycles (Cycles 2, 4, and 6), and methotrexate, 1000 mg/m^2 (<60 yrs) and 250 mg/m^2 (≥60 yrs), IV infusion, on Day 1 of each 28-day odd cycles (Cycle 1, 3, and 5) in consolidation phase followed by imatinib 600 mg, tablets, orally, QD, along with vincristine 1.4 mg/m^2 (max 2 mg), IV, on Day 1 and prednisone 200 mg (<60 yrs), 100 mg (≥60-69 yrs) and 50 mg (≥70 yrs) on Days 1 through 5 in each 28-day cycle up to 11 cycles in maintenance phase up to data cut-off date: 12 August 2022.
  Interventions: Drug: Imatinib; Drug: Vincristine; Drug: Dexamethasone; Drug: Cytarabine; Drug: Methotrexate; Drug: Prednisone

INTERVENTIONS:
Drug: Ponatinib — Ponatinib Tablets.
  Other Names: Iclusig
  Arms: Cohort A: Ponatinib 30 milligram (mg)
Drug: Imatinib — Imatinib Tablets.
  Other Names: Gleevec
  Arms: Cohort B: Imatinib 600 mg
Drug: Vincristine — Vincristine IV injection.
Drug: Dexamethasone — Dexamethasone Tablets.
Drug: Cytarabine — Cytarabine IV infusion.
Drug: Methotrexate — Methotrexate IV infusion.
Drug: Prednisone — Prednisone Tablets.

SUMMARY:
In this study, adults with newly-diagnosed Philadelphia Chromosome-positive acute lymphoblastic leukemia (Ph+ ALL) will receive first-line therapy of ponatinib or imatinib.

The main aim of this study is to compare the number of participants on each treatment that show no signs of disease.

Participants will take tablets of either ponatinib or imatinib at the same time each day combined with reduced-intensity chemotherapy for up to 20 months. Then, they will continue with single-agent therapy (ponatinib or imatinib) until they meet the discontinuation criteria from the study.

DETAILED DESCRIPTION:
The drug being tested in this study is called ponatinib. Ponatinib is being tested to treat people who have newly diagnosed Ph+ ALL. This study will look at the efficacy of ponatinib in participants in addition to standard care.

The study will enroll approximately 230 participants. Participants will be randomized in a 2:1 ratio to receive oral ponatinib or imatinib (Cohort A and Cohort B, respectively) daily throughout the study.

All participants will be asked to take ponatinib or imatinib at the same time each day with reduced-intensity chemotherapy in induction phase (Cycles 1 to 3), consolidation phase (Cycles 4 to 9) and maintenance phase (Cycles 10 to 20). At the end of the 20 cycles, participants will remain on ponatinib or imatinib (administered as a single agent). The dose of ponatinib in consolidation and maintenance phase will start with the last dose given in the previous phase. The dose can be modified based on MRD-negative CR results.

This multi-center trial will be conducted in Argentina, Australia, Austria, Belarus, Brazil, Bulgaria, Canada, Chile, France, Mexico, Greece, Italy, Japan, Korea, Republic Of, Poland, Romania, Russia, Spain, Taiwan, Province Of China, Turkey, Finland and the United States. Participants including those who achieve a clinical response, may receive study drug until they are deceased, have failed to achieve the primary endpoint, have experienced relapse from CR or have progressive disease, have an unacceptable toxicity, have withdrawn consent, have proceeded to HSCT, or until the sponsor terminates the study, whichever occurs first. After disease progression, all participants will be contacted every 3 months for survival follow-up. Participants will be followed until completion of the study or until the participant's death has been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Philadelphia chromosome-positive (Ph+) or BCR-ABL1-positive ALL, as defined by the 2017 national comprehensive cancer network (NCCN) guidelines.
2. Eastern Cooperative Oncology Group (ECOG) performance status of <=2.

Exclusion Criteria:

1. With a history or current diagnosis of chronic phase, accelerated phase, or blast phase chronic myeloid leukemia (CML).
2. Prior/current treatment with any systemic anticancer therapy (including but not limited to any tyrosine kinase inhibitor [TKI]) and/or radiotherapy for ALL, with the exception of an optional prephase therapy or chemotherapy induction (no more than 1 cycle), which should be discussed with the sponsor's medical monitor/designee.
3. Currently taking drugs that are known to have a risk of causing prolonged corrected QT (QTc) or torsades de pointes (TdP) (unless these can be changed to acceptable alternatives or discontinued).
4. Taking any medications or herbal supplements that are known to be strong inhibitors or strong inducers of cytochrome P450 (CYP)3A4 within at least 14 days before the first dose of study drug.
5. Uncontrolled active serious infection that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
6. Major surgery within 28 days before randomization (minor surgical procedures such as catheter placement or BM biopsy are not exclusionary criteria).
7. Known human immunodeficiency virus (HIV) seropositivity, known active hepatitis B or C infection.
8. History of acute pancreatitis within 1 year of study screening or history of chronic pancreatitis.
9. Uncontrolled hypertriglyceridemia (triglycerides >450 milligram per deciliter [mg/dL]).
10. Diagnosed and treated for another malignancy within 5 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
11. History or presence of clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
12. Clinical manifestations of CNS or extramedullary involvement with ALL other than lymphadenopathy or hepatosplenomegaly.
13. Autoimmune disease with potential CNS involvement.
14. Known significant neuropathy of Grade >=2 severity.
15. Clinically significant, uncontrolled, or active cardiovascular, cerebrovascular, or peripheral vascular disease, or history of or active venous thrombotic/embolic event (VTE) disease.
16. Have a significant bleeding disorder unrelated to ALL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2027-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (92):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope - Duarte, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Indiana Blood & Marrow Transplantation, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center, New Hyde Park, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Oregon Health and Science University, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
- Argentina (2):
  - Sanatorio Allende, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
- Australia (3):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
- Austria (3):
  - Ordensklinikum Linz Elisabethinen, Linz, Upper Austria
  - Hanusch Krankenhaus Wiener Gebietskrankenkasse, Vienna, Vienna
  - Universitaetsklinik Fuer Innere Medizin I, Vienna
- Brazil (10):
  - Hospital Sao Rafael-Monte Tabor, Salvador, Estado de Bahia
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital da Cidade, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hemocentro Campinas Unicamp, Campinas, São Paulo
  - Fundacao Doutor Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Riberao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - HEMORIO Instituto Estadual de Hematologia Arthur Siqueira de Cavalcanti, Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente - A.C.Camargo Cancer Center, São Paulo
- University Multiprofile Hospital for Active Treatment Saint Ivan Rilski, Sofia, Sofia, Bulgaria
- Canada (4):
  - 855 West 12th Avenue, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital Charles-LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- China (5):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Soochow University/Suzhou First People's Hospital, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Institute of Hematology & Blood Diseases Hospital of CAMS & PUMC, Tianjin
- Helsingin ja Uudenmaan sairaanhoitopiiri, Helsinki, Finland
- France (4):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse, Midi-pyrenees
  - Center Hospitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Centre Hospitalier de Versailles Hopital Andre Mignot, Le Chesnay, Île-de-France Region
- Greece (3):
  - University General Hospital of Athens Attikon, Chaïdári, Attica
  - Evaggelismos General Hospital, Athens, Ipsiladou 45-47
  - General University Hospital of Patras Panagia I Voithia, Pátrai, Rio
- Italy (13):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-cesena
  - Azienda Policlinico San Martino, Genoa, Liguria
  - Azienda Ospedaliera San Gerardo di Monza, Monza, Monza E Brianza
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Reggio Nella Emilia
  - Ospedale dell'Angelo, Mestre, Venezia
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Istituto Scientifico Universitario San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria di Modena Policlinico, Modena
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Azienda USL della Romagna, Ravenna
  - Centro di Ematologia Policlinico Umberto I Universita Sapienza di Roma, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Japan (6):
  - Chiba Aoba Municipal Hospital, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Aiiku Hospital, Sapporo, Hokkaido
  - Tokai University Hospital, Isehara, Kanagawa
  - Okayama University Hospital, Okayama, Okayama-ken
- Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León, Mexico
- Poland (4):
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych z Warminsko-Mazurs, Olsztyn, Warmian-Masurian Voivodeship
- Russia (4):
  - City Clinical Hospital named after Vikentiy Vikentyevich Veresaev, Moscow, Moscow CITY
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg, Sverdlovsk Oblast
  - National Research Center for Hematology, Dept. of Hematology/Oncology and BMT, Moscow
  - Almazov Federal North-West Medical Research Centre of Department of Health of Russian Federation, Saint Petersburg
- South Korea (5):
  - The Catholic University of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Hospital, Daegu
- Spain (4):
  - Institut Catala d'Oncologia Badalona - Hospital Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (3):
  - Hualien Tzu Chi Hospital, Hualien City, Hualien
  - China Medical University Hospital, Taichung, Taichung CITY
  - National Cheng Kung University Hospital, Tainan, Tainan CITY
- Ankara Universitesi Tp Fakultesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ashaye A, Shi L, Aldoss I, Montesinos P, Vachhani P, Rocha V, Papayannidis C, Leonard JT, Baer MR, Ribera JM, McCloskey J, Wang J, Rane D, Guo S. Quality-Adjusted Time Without Symptoms of Disease or Toxicity (Q-TWiST) in Patients With Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia: A Comparison of Ponatinib Versus Imatinib. Cancer Med. 2025 Apr;14(7):e70780. doi: 10.1002/cam4.70780. PMID 40165400
- [Derived] Jabbour E, Kantarjian HM, Aldoss I, Montesinos P, Leonard JT, Gomez-Almaguer D, Baer MR, Gambacorti-Passerini C, McCloskey J, Minami Y, Papayannidis C, Rocha V, Rousselot P, Vachhani P, Wang ES, Wang B, Hennessy M, Vorog A, Patel N, Yeh T, Ribera JM. Ponatinib vs Imatinib in Frontline Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia: A Randomized Clinical Trial. JAMA. 2024 Jun 4;331(21):1814-1823. doi: 10.1001/jama.2024.4783. PMID 38722621

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 77 investigative sites in Australia, China, Korea, Taiwan, Austria, France, Greece, Italy, Poland, Russia, Spain, Turkey, United States, Canada, Mexico, Argentina and Brazil from 04 October 2018 to 31 July 2027. This study is ongoing. The data is reported for primary outcome measures up to 12 August 2022.
Pre-assignment Details: Participants with a diagnosis of Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL) were enrolled in a 2:1 ratio to receive ponatinib or imatinib.
Groups:
- Cohort A: Ponatinib 30 mg: Ponatinib 30 mg, tablets, orally, once daily (QD), with vincristine 1.4 mg/m^2 (max 2 mg) intravenous (IV), on Days 1 and 14 and dexamethasone 40 mg (<60 years [yrs]) and 20 mg (≥60 yrs), orally, once on Days 1 to 4, Days 11 to 14 for up to 3 cycles (each cycle=28 days) in induction phase (IP) (reduced dose of ponatinib 15 mg upon achievement of MRD-negative CR at end of induction) followed by ponatinib last induction phase dose with cytarabine, 1000 mg/m^2 as 2-hour IV infusion (<60 yrs) and 250 mg/m^2 (≥60 yrs) every 12 hours, IV on Days 1, 3, 5 of Cycles 2,4,6 and methotrexate, 1000 mg/m^2 (<60 yrs) and 250 mg/m^2 (≥60 yrs), IV infusion, on Day 1 of cycles 1, 3, 5 in consolidation phase (CP) followed by ponatinib last consolidation phase dose with vincristine 1.4 mg/m^2 (max 2 mg), IV, on Day 1 and prednisone 200 mg (<60 yrs), 100 mg (≥60-69 yrs) and 50 mg(≥70 yrs) on Days 1 to 5 for up to 11 cycles in maintenance phase (MP) up to data cut-off date: 12 August 2022.
Period: IP (Cycles 1-3) (Cycle Length=28 Days)
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Imatinib 600 mg
Started | 164 | 81
Efficacy Evaluable Population (Efficacy evaluable population was defined as all participants in the ITT population with BCR:ABL1 dominant variant of p190 or p210 confirmed by central lab.) | 154 | 78
Safety Population (The safety population was defined as all participants who were randomized to the ponatinib or imatinib arm and received at least 1 dose of any study drug.) | 163 | 81
Completed | 0 | 0
Not Completed | 164 | 81
Not completed — Participants Ongoing on Study | 135 | 63
Not completed — Death | 21 | 13
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Reason not Specified | 2 | 0
Period: CP (Cycles 4-9) (Cycle Length=28 Days)
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Imatinib 600 mg
Started (Participants are still ongoing in Induction Phase.) | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: MP (Cycles 10-20) (Cycle Length=28 Days)
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Imatinib 600 mg
Started (Participants are still ongoing in Induction Phase.) | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis set was defined as all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Imatinib 600 mg | Total
Number analyzed (Participants) | 164 | 81 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (16.09) | 50.6 (14.60) | 51.0 (15.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 43 | 133
  Male | 74 | 38 | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 20 | 11 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 4 | 13
  White | 104 | 62 | 166
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 28 | 2 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 20 | 59
  Non-Hispanic and Latino | 105 | 56 | 161
  Not reported | 15 | 4 | 19
  Unknown | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 4 | 2 | 6
  China | 14 | 8 | 22
  Korea, South | 1 | 2 | 3
  Taiwan | 3 | 0 | 3
  Austria | 3 | 3 | 6
  France | 9 | 1 | 10
  Greece | 4 | 1 | 5
  Italy | 28 | 10 | 38
  Poland | 5 | 2 | 7
  Russia | 5 | 6 | 11
  Spain | 16 | 9 | 25
  Turkey | 1 | 1 | 2
  Canada | 8 | 5 | 13
  Mexico | 2 | 1 | 3
  United States | 40 | 20 | 60
  Argentina | 3 | 0 | 3
  Brazil | 18 | 10 | 28
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number analyzed are the number of participants available for height at baseline.
  centimeters (cm)
    number analyzed (Participants) | 158 | 76 | 234
    (all) | 167.24 (9.980) | 167.27 (9.029) | 167.25 (9.662)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number analyzed are the number of participants available for weight at baseline.
  kilograms (kg)
    number analyzed (Participants) | 163 | 81 | 244
    (all) | 74.17 (18.675) | 76.23 (18.565) | 74.86 (18.626)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: meters squared (m^2)] — Population: Number analyzed are the number of participants available for BSA at baseline.
  meters squared (m^2)
    number analyzed (Participants) | 157 | 76 | 233
    (all) | 1.84 (0.261) | 1.86 (0.255) | 1.85 (0.258)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Minimal Residual Disease (MRD)-Negative Complete Remission (CR) at The End of Induction Phase
Description: MRD-negative CR was achieved when a participant met the criteria for both MRD negativity and CR. MRD-negativity: ≤0.01 % breakpoint cluster region-Abelson (BCR-ABL1/ABL1), or undetectable BCR-ABL1 transcripts in complementary deoxyribonucleic acid (cDNA) with ≥ 10,000 ABL1 transcripts. CR: meeting all the following for at least 4 weeks (that is no recurrence):1. No circulating blasts and less than (<) 5% blasts in the bone marrow (BM). 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (central nervous system [CNS] involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. Absolute neutrophil count (ANC) > 1000 per microliter (/mcL) (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L).
Time Frame: From Cycle 1 through Cycle 3 (approximately 3 months) (Cycle length = 28 days)
Population: ITT population with p190/p210 variant was defined as all participants in the ITT population who were identified by the central laboratory as having baseline breakpoint cluster region-Abelson1 (BCR-ABL1) dominant variants of p190 or p210.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Imatinib 600 mg
Number analyzed (Participants) | 154 | 78
Participants | 53 | 13
Statistical Analysis 1: Comparison: Cohort A: Ponatinib 30 mg vs Cohort B: Imatinib 600 mg; Test type: Superiority; p = 0.0021, Chi-squared — P-value is based on CMH chi-square test, with stratification according to randomization strata (age): 18 through <45 years, ≥45 through <60 years, and ≥60 years; Risk Difference (RD) = 0.18, 95% CI 2-sided [0.06 to 0.29] — Risk difference and 95% CI: adjusted percent ponatinib - adjusted percent imatinib and its 95% CI

2. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the dates of randomization until death due to any cause or failure to achieve CR by end of induction or relapse from CR. CR: meeting all the following for at least 4 weeks (that is no recurrence):1. No circulating blasts and less than (<) 5% blasts in the bone marrow (BM). 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (central nervous system [CNS] involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. Absolute neutrophil count (ANC) greater than (>) 1000 per micro liter (/mcL) (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L).Relapse from CR: reappearance of blasts in the blood or BM (>=5%) or in any extramedullary site after a CR.
Time Frame: Baseline up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

3. Secondary Outcome: Percentage of Participants With CR and Incomplete Complete Remission (CRi)
Description: CR is defined as meeting all the following for at least 4 weeks (that is, no recurrence): 1. No circulating blasts and <5% blasts in the BM. 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (CNS involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. ANC >1000/mcL (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L). CRi is defined as hematologic complete remission with incomplete hematologic recovery and meeting all criteria for CR except platelet count and/or ANC.
Time Frame: End of Cycle 1 (approximately 1 month), Cycle 2 (approximately 2 months), Cycle 3 (approximately 3 months), and Cycle 9 (approximately 9 months) (Cycle length= 28 days)
Reporting Status: Not Posted, anticipated posting 2028-07

4. Secondary Outcome: Percentage of Participants With Molecular Response
Description: Molecule response is assessed by 3-Log Reduction (MR3), Molecular Response 4-Log Reduction (MR4) and Molecular Response 4.5-Log Reduction (MR4.5). MR3 is defined as molecular response 3-log reduction (<=0.1% BCR-ABL1/ABL1), or undetectable BCR-ABL1 transcripts in cDNA with >=1000 ABL1 transcripts. MR4 is defined as molecular response 4-log reduction (<=0.01% BCR-ABL1/ABL1), or undetectable BCR-ABL1 transcripts in cDNA with >=10,000 ABL1 transcripts. MR4.5 is defined as Molecular response 4.5-log reduction (<=0.0032% BCR-ABL1/ABL1), or undetectable BCR-ABL1 transcripts in cDNA with >=32,000 ABL1 transcripts.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2028-07

5. Secondary Outcome: Percentage of Participants With Primary Induction Failure (PIF)
Description: PIF is defined as participants who received treatment for ALL but never achieved CR or CRi by the end of induction. PIF is not limited by the number of unsuccessful treatments; this disease status only applies to recipients who have never been in CR or CRi. CR is defined as meeting all the following for at least 4 weeks (that is no recurrence): 1. No circulating blasts and <5% blasts in the BM. 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (CNS involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. ANC >1000/mcL (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L). CRi is defined as hematologic complete remission with incomplete hematologic recovery and meeting all criteria for CR except platelet count and/or ANC.
Time Frame: Up to 3 months
Reporting Status: Not Posted, anticipated posting 2028-07

6. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR is defined as CR + CRi by end of induction. CR is defined as meeting all the following for at least 4 weeks (that is no recurrence): 1. No circulating blasts and <5% blasts in the BM. 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (CNS involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. ANC >1000/mcL (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L). CRi is defined as hematologic complete remission with incomplete hematologic recovery and meeting all criteria for CR except platelet count and/or ANC.
Time Frame: Up to 3 months
Reporting Status: Not Posted, anticipated posting 2028-07

7. Secondary Outcome: Percentage of MRD-Negative CR
Description: MRD is defined as the percentage of participants achieving CR who are MRD-negative at multiple intervals after end of induction. MRD negativity: <=0.01% BCR-ABL1/ABL1, or undetectable BCR-ABL1 transcripts in cDNA with >=10,000 ABL1 transcripts. Relapse from CR: Reappearance of blasts in the blood or BM (>=5%) or in any extramedullary site after a CR.
Time Frame: Up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

8. Secondary Outcome: Duration of MRD-Negative CR
Description: Duration of MRD-negative CR is defined as interval between the first assessment at which the criteria for MRD-negative CR are met until the earliest date at which loss of MRD negativity or relapse from CR occurs. MRD negativity (MR4): <=0.01% BCR-ABL1/ABL1, or undetectable BCR-ABL1 transcripts in cDNA with >=10,000 ABL1 transcripts. CR is defined as meeting all the following for at least 4 weeks (that is, no recurrence): 1. No circulating blasts and <5% blasts in the BM. 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (CNS involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. ANC >1000/mcL (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L). Relapse from CR: Reappearance of blasts in the blood or BM (>=5%) or in any extramedullary site after a CR.
Time Frame: Up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

9. Secondary Outcome: Duration of CR
Description: Duration of CR is defined as interval between the first assessment at which the criteria for CR are met until the earliest date at which relapse from CR occurs. CR is defined as meeting all the following for at least 4 weeks (that is no recurrence): 1. No circulating blasts and <5% blasts in the BM. 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (CNS involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. ANC >1000/mcL (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L). Relapse from CR: Reappearance of blasts in the blood or BM (>=5%) or in any extramedullary site after a CR.
Time Frame: Up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

10. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as time to end of study randomized treatment (except for hematopoietic stem cell transplantation [HSCT] without loss of MRD-negative CR) due to safety and efficacy reasons. MRD-negative CR is achieved when a participant meets the criteria for both MRD negativity and CR. MRD-negativity: <=0.01% BCR-ABL1/ABL1, or undetectable BCR-ABL1 transcripts in cDNA with >=10,000 ABL1 transcripts. CR: meeting all the following for at least 4 weeks (that is no recurrence):1. No circulating blasts and <5% blasts in the BM. 2. Normal maturation of all cellular components in the BM. 3. No extramedullary disease (CNS involvement, lymphadenopathy, splenomegaly, skin/gum infiltration, testicular mass). 4. ANC >1000/mcL (or >1.0*10^9/L). 5. Platelets >100,000/mcL (or >100*10^9/L).
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

11. Secondary Outcome: Duration of MR4.5
Description: Duration of MR4.5 is defined as interval between the first assessment at which the criteria for MR4.5 are met until the earliest date at which loss of MR4.5 occurs. MR4.5 is molecular response 4.5-log reduction (<=0.0032% BCR-ABL1/ABL1), or undetectable BCR-ABL1 transcripts in cDNA with >=32,000 ABL1 transcripts.
Time Frame: Up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

12. Secondary Outcome: Percentage of On-Study Participants With Overall Survival (OS)
Description: On-study participants with or without HSCT will be evaluated. OS is defined as interval between randomization and death due to any cause, censored at the last contact date when the participant was alive.
Time Frame: Up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

13. Secondary Outcome: Percentage of On-Study Participants With Relapse From CR
Description: On-study participants with or without HSCT will be evaluated. Relapse from CR is defined as reappearance of blasts in the blood or BM (>=5%) or in any extramedullary site after a CR.
Time Frame: Up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

14. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as interval between the randomization and death due to any cause, censored at the last contact date when the participant was alive.
Time Frame: Up to approximately 3 to 6 years
Reporting Status: Not Posted, anticipated posting 2028-07

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to data cut-off date: 12 August 2022 (up to 46 months 1 week)
Description: Safety population was defined as all participants who were randomized to the ponatinib or imatinib arm and received at least 1 dose of any study drug.
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Imatinib 600 mg
All-Cause Mortality (participants affected / at risk) | 21/163 | 13/81
Serious Adverse Events (participants affected / at risk) | 97/163 | 45/81
Other Adverse Events (participants affected / at risk) | 159/163 | 80/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ponatinib 30 mg (N=163) | Cohort B: Imatinib 600 mg (N=81)
Septic shock (Infections and infestations) | 6 | 3
COVID-19 (Infections and infestations) | 7 | 1
Sepsis (Infections and infestations) | 6 | 2
Pneumonia (Infections and infestations) | 4 | 3
COVID-19 pneumonia (Infections and infestations) | 3 | 2
Cellulitis (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Klebsiella sepsis (Infections and infestations) | 2 | 0
Vascular device infection (Infections and infestations) | 2 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Mucormycosis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
SARS-CoV-2 viraemia (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Stenotrophomonas bacteraemia (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 27 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 0
Ataxia (Nervous system disorders) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 3
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Platelet count decreased (Investigations) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin unconjugated increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
pH urine decreased (Investigations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Brachiocephalic vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Psychomotor retardation (Psychiatric disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Immunisation reaction (Immune system disorders) | 1 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ponatinib 30 mg (N=163) | Cohort B: Imatinib 600 mg (N=81)
Alanine aminotransferase increased (Investigations) | 67 | 27
Lipase increased (Investigations) | 44 | 29
Platelet count decreased (Investigations) | 39 | 26
Neutrophil count decreased (Investigations) | 34 | 26
Aspartate aminotransferase increased (Investigations) | 39 | 15
White blood cell count decreased (Investigations) | 25 | 20
Gamma-glutamyltransferase increased (Investigations) | 21 | 8
Blood lactate dehydrogenase increased (Investigations) | 19 | 8
Amylase increased (Investigations) | 16 | 10
Blood alkaline phosphatase increased (Investigations) | 14 | 7
Blood creatinine increased (Investigations) | 10 | 8
Blood bilirubin increased (Investigations) | 14 | 3
Blood fibrinogen decreased (Investigations) | 9 | 5
C-reactive protein increased (Investigations) | 8 | 5
Lymphocyte count decreased (Investigations) | 5 | 8
Weight decreased (Investigations) | 7 | 6
Transaminases increased (Investigations) | 10 | 2
Nausea (Gastrointestinal disorders) | 57 | 40
Constipation (Gastrointestinal disorders) | 62 | 17
Vomiting (Gastrointestinal disorders) | 36 | 31
Diarrhoea (Gastrointestinal disorders) | 28 | 26
Stomatitis (Gastrointestinal disorders) | 31 | 15
Abdominal pain (Gastrointestinal disorders) | 25 | 10
Abdominal pain upper (Gastrointestinal disorders) | 23 | 6
Dyspepsia (Gastrointestinal disorders) | 14 | 7
Haemorrhoids (Gastrointestinal disorders) | 15 | 4
Toothache (Gastrointestinal disorders) | 10 | 3
Abdominal distension (Gastrointestinal disorders) | 9 | 3
Anaemia (Blood and lymphatic system disorders) | 71 | 44
Thrombocytopenia (Blood and lymphatic system disorders) | 75 | 31
Neutropenia (Blood and lymphatic system disorders) | 70 | 30
Leukopenia (Blood and lymphatic system disorders) | 23 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 18 | 7
Leukocytosis (Blood and lymphatic system disorders) | 16 | 4
Headache (Nervous system disorders) | 69 | 35
Neuropathy peripheral (Nervous system disorders) | 51 | 19
Paraesthesia (Nervous system disorders) | 33 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 18 | 10
Dizziness (Nervous system disorders) | 16 | 10
Hypoaesthesia (Nervous system disorders) | 10 | 1
Dysgeusia (Nervous system disorders) | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 40 | 31
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 22 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 17 | 17
Decreased appetite (Metabolism and nutrition disorders) | 15 | 15
Hyperuricaemia (Metabolism and nutrition disorders) | 16 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | 9
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 8
Pyrexia (General disorders) | 57 | 19
Fatigue (General disorders) | 43 | 18
Oedema peripheral (General disorders) | 17 | 26
Asthenia (General disorders) | 26 | 12
Pain (General disorders) | 10 | 4
Chest pain (General disorders) | 11 | 1
Face oedema (General disorders) | 3 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 12 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 6
Hypertension (Vascular disorders) | 52 | 11
Hypotension (Vascular disorders) | 10 | 4
Deep vein thrombosis (Vascular disorders) | 8 | 5
Rash (Skin and subcutaneous tissue disorders) | 31 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 9 | 2
COVID-19 (Infections and infestations) | 21 | 7
Urinary tract infection (Infections and infestations) | 13 | 2
Conjunctivitis (Infections and infestations) | 12 | 2
Pneumonia (Infections and infestations) | 10 | 2
Folliculitis (Infections and infestations) | 9 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Insomnia (Psychiatric disorders) | 31 | 14
Anxiety (Psychiatric disorders) | 14 | 7
Depression (Psychiatric disorders) | 9 | 5
Vision blurred (Eye disorders) | 12 | 3
Periorbital oedema (Eye disorders) | 1 | 7
Tachycardia (Cardiac disorders) | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03589326/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03589326/SAP_001.pdf